CLINICAL TRIAL: NCT05727163
Title: FOLFOX Via Hepatic Artery Infusion Chemotherapy (HAI) Plus Systemic Irinotecan With or Without Bevacizumab Versus Systemic FOLFOXIRI With or Without Bevacizumab in Patients With Initially Unresectable RAS-mutated Colorectal Cancer With Liver Metastases: A Prospective, Randomized, Controlled Clinical Study
Brief Title: FOLFOX Via HAI Plus Intravenous Irinotecan With or Without Bevacizumab Versus Systemic FOLFOXIRI With or Without Bevacizumab in Initially Unresectable RAS-mutated CRLM Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: New Triumph
Record Dates: First submitted 2022-10-24; First posted 2023-02-14 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal liver metastasis; Hepatic Artery Infusion Chemotherapy; RAS-mutation; Systemic Chemotherapy; FOLFOX; FOLFOXIRI; Initially unresectable colon cancer
MeSH Terms: interventions — Dexamethasone; anisodamine; 2-(phenylmethyl)-1-naphthol; Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAI group (Experimental): FOLFOX given via Hepatic Artery Infusion (HAI) in Combination With intravenous Irinotecan With or Without Bevacizumab.
  Dexamethasone 25 mg via HAI (Pre-chemotherapy) Anisodamine (654-2) 10 mg HAI (Pre-chemotherapy) Oxaliplatin 85 mg/m2 via HAI over 3 hours Leucovorin 200 mg/m2 via HAI FU 400 mg/m2 via HAI FU 2.4g/m2 via HAI over 48 hours Irinotecan 150 mg/m2 intravenously Bevacizumab 5 mg/kg intravenously
  The above regimen was given on Day 1 and repeated after 14 days. Patients will typically receive a maximum of 12 courses (preoperative and/or postoperative) unless disease progression is detected, intolerable adverse effects, or the patient refuses further treatment.
  Interventions: Drug: Dexamethasone; Drug: Anisodamine; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Irinotecan; Drug: Bevacizumab
- Systemic Chemotherapy group (Active Comparator): Systemic FOLFOXIRI With or Without Bevacizumab
  Irinotecan 150mg/m2 intravenously Oxaliplatin 85 mg/m2 intravenously over 3 hours Leucovorin 200 mg/m2 intravenously FU 400 mg/m2 intravenously 5-FU 2400 mg/m2 continuous intravenous infusion over 46 hours Bevacizumab 5 mg/kg intravenously
  Note: (UGT*28 7/7, UGT*6 A/A, UGT*28 6/7 and UGT*6 A/G patients, Irinotecan dosage was reduced to 130 mg/m2)
  The above regimen was given on Day 1 and repeated after 14 days. Patients will typically receive a maximum of 12 courses (preoperative and/or postoperative) unless disease progression is detected, intolerable adverse effects, or the patient refuses further treatment.
  Interventions: Drug: Irinotecan; Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Dexamethasone — 25mg via HAI (Pre-chemotherapy)
  Arms: HAI group
Drug: Anisodamine — 10 mg via HAI (Pre-chemotherapy)
  Other Names: 654-2
  Arms: HAI group
Drug: Oxaliplatin — 85 mg/m2 via HAI over 3 hours
  Arms: HAI group
Drug: Leucovorin — 200 mg/m2 via HAI
  Arms: HAI group
Drug: Fluorouracil — 400 mg/m2 via HAI and 2.4g/m2 via HAI over 48 hours
  Other Names: FU
  Arms: HAI group
Drug: Irinotecan — 150 mg/m2 intravenously
Drug: Bevacizumab — 5 mg/kg intravenously
Drug: Oxaliplatin — 85 mg/m2 intravenously over 3 hours
  Arms: Systemic Chemotherapy group
Drug: Leucovorin — 200 mg/m2 intravenously
  Arms: Systemic Chemotherapy group
Drug: Fluorouracil — 400 mg/m2 intravenously + 2400 mg/m2 continuous intravenous infusion over 46 hours
  Other Names: FU
  Arms: Systemic Chemotherapy group

SUMMARY:
This prospective, randomized, controlled clinical study aims to evaluate the objective remission rate of FOLFOX hepatic artery infusion chemotherapy (HAI) in combination with systemic irinotecan with or without bevacizumab versus systemic intravenous FOLFOXIRI with or without bevacizumab in initially unresectable RAS-mutated colorectal cancer patients with liver metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

The goal of this prospective, randomized, controlled clinical trial is to evaluate the objective remission rate (ORR) of FOLFOX hepatic artery infusion chemotherapy (HAI) in combination with irinotecan with or without bevacizumab systemic intravenous chemotherapy versus systemic intravenous FOLFOXIRI with or without bevacizumab in initially unresectable RAS-mutated colorectal cancer patients with liver metastases.

SECONDARY OBJECTIVES:

To assess and compare the depth of response (DpR), R0 surgical resection rate, No evidence of disease (NED) rate, progression-free survival (PFS), overall survival (OS), recurrence-free survival (RFS) in resectable patients and safety (chemotherapy-related adverse events, catheterization-related adverse events, surgical complications, etc.) between the two intervention groups.

OUTLINE:

Patients in the HAI group receive FOLFOX via hepatic artery infusion chemotherapy plus intravenous irinotecan with or without bevacizumab every 14 days, while patients in the systemic group receive intravenous FOLFOXIRI regimen with or without bevacizumab every 14 days. Patients will receive a maximum of 12 cycles in total (before and after surgery) unless there is disease progression, unacceptable toxicity, or if the patient withdraws from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal adenocarcinoma
2. Imaging or pathological confirmation of liver metastases
3. The multidisciplinary team determined that the liver metastases were unresectable, defined as (i) ≥5 metastases; (ii) inability to perform R0 resection; (iii) insufficient volume of liver expected to remain after resection; (iv) failure to preserve all 3 hepatic veins after resection, failure to ensure that blood flow to and from the liver and bile ducts can be preserved, and failure to preserve 2 adjacent liver segments. If any of the above criteria are met, it can be considered as initially unresectable liver metastases.
4. Patients with mutated RAS and BrafV600E
5. No previous treatment for liver metastases, including chemotherapy, surgery, radiotherapy, transarterial chemoembolization (TACE) and targeted therapy
6. No extrahepatic metastases confirmed by CT, MRI, or PET/CT (if necessary) (consider enrollment if there is a lung or lymph node lesion less than 10 mm and metastases are difficult to identify)
7. Normal hematological function (platelets >90×109/L; white blood cells >3×109/L; neutrophils >1.5×109/L)
8. Serum bilirubin ≤ 1.5 times the upper limit of normal value (ULN), transaminases ≤ 5 times ULN
9. No ascites, normal coagulation function, albumin ≥35g/L
10. Liver function Child-Push grade A
11. Serum creatinine less than upper limit of normal (ULN) or calculated creatinine clearance >50 ml/min (using Cockcroft-Gault formula)
12. ECOG score 0-1
13. Life expectancy > 3 months
14. Signed written informed consent

Exclusion Criteria (Patients meeting any of the following criteria will be excluded from the study):

1. Presence of any extrahepatic metastases and/or primary tumor not amenable to radical surgical resection
2. Development of liver metastases within 1 year after completion of adjuvant chemotherapy with FOLFOX or XELOX
3. Severe arterial embolism or ascites
4. Bleeding tendency or coagulation disorder
5. Hypertensive crisis or hypertensive encephalopathy
6. Severe uncontrolled systemic complications such as infections or diabetes mellitus
7. Clinically significant cardiovascular disease such as cerebrovascular accident (within 6 months prior to enrollment), myocardial infarction (within 6 months prior to enrollment), uncontrolled hypertension despite appropriate medication, unstable angina pectoris, congestive heart failure (NYHA class 2-4), arrhythmias requiring medication
8. History or physical examination revealing a central nervous system disease (e.g., primary brain tumor, epilepsy not manageable by standard therapy, presence of brain metastases, or history of stroke)
9. Previous malignancy within the last 5 years (except post-radical surgery basal cell carcinoma of the skin and/or carcinoma in situ of the cervix)
10. Treatment using any investigational drug within the last 28 days prior to the study
11. Any residual toxicity from prior chemotherapy (except alopecia), such as peripheral neuropathy ≥ NCI CTC v3.0 grade 2, will not be considered for treatment with oxaliplatin-containing regimens
12. History of allergy to any of the drugs in the study
13. Women of childbearing potential (<2 years after last menstruation) or men of childbearing potential who are not using or have refused to use an effective non-hormonal contraceptive (IUD, barrier method combined with spermicidal gel or sterilization) during pregnancy and lactation
14. Unable or unwilling to comply with the study protocol
15. Presence of any other disease, dysfunction due to metastatic lesions, or suspicious medical findings that suggest a possible contraindication to the use of the study drug or that would place the patient at risk of treatment-related complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Remission Rate (ORR) | Assessed up to 48 months
  As assessed by the investigators using RECIST v1.1 criteria

SECONDARY OUTCOMES:
Depth of Response (DpR) | Assessed up to 48 months
  The investigators evaluate the maximum tumor regression to baseline tumor ratio to determine the depth of tumor regression (DpR) and calculate the median value.
R0 surgical resection rate | Assessed up to 48 months
  Defined as the proportion of patients who achieved complete resection (pathologically determined R0 resection) after treatment
No evidence of disease rate (NED) | Assessed up to 48 months
  Proportion of treated patients who achieve no evidence of disease
Progression Free Survival (PFS) | Assessed up to 48 months
  The length of time during and after the treatment of the disease, that a patient lives with the disease without its aggravation
Overall Survival (OS) | Assessed up to 48 months
  The length of time from the start of treatment that patients diagnosed are still alive
Recurrence Free Survival in resectable patients | Assessed up to 48 months
  Defined as the time from complete resection of liver metastases or NED to the development of disease recurrence or death
Safety (including chemotherapy-related adverse events, catheterization-related adverse events, surgical complications, etc.) | Assessed up to 48 months
  Number of patients with adverse events and severity according to NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided